CLINICAL TRIAL: NCT03341364
Title: Acceptance and Commitment Based Group Therapy for Cancer Patients: a Pilot Study Comparing ACT-group Therapy With Individual ACT Therapy for Cancer Patients Experiencing Psychological Distress
Brief Title: Acceptance and Commitment Based Group Therapy for Cancer Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Central contact person ended employment
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2017/602
Record Dates: First submitted 2017-10-25; First posted 2017-11-14 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Cancer; Psychological Distress
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Recruitment of participants to the group intervention will start first. When a maximum of 10 participants have been recruited to the group intervention and/or one week before start of group intervention, recruitment to the Active Control group will start. The individual therapies will start at different times, depending on the flow of referrals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT group treatment (Experimental): Participants receiving the ACT-based group therapy.
  Interventions: Behavioral: ACT-based group therapy
- ACT individual (Active Comparator): Participants receiving individual ACT-based therapy.
  Interventions: Behavioral: ACT individual treatment

INTERVENTIONS:
Behavioral: ACT-based group therapy — 6 group therapy sessions over 6 weeks (one session à 2 hours weekly), plus one follow-up session 6 weeks after last session. The sessions are lead by a psychologist and a social worker. Each session containing discussions, experimental exercises and home-work assignment.
  Arms: ACT group treatment
Behavioral: ACT individual treatment — 3-12 individual therapy sessions over 3-16 weeks, plus one follow-up session 6 weeks after last session, lead by a clinical psychologist. Each session containing discussion, experimental exercises and home-work assignment.
  Arms: ACT individual

SUMMARY:
This study evaluates the preliminary effects of an Acceptance and Commitment (ACT)-based group therapy compared to individual ACT-therapy for adult cancer patients suffering from psychological distress. Half of the participants will receive ACT in a group setting, while the other half will receive individual ACT.

DETAILED DESCRIPTION:
This study evaluates the preliminary effects of an Acceptance and Commitment (ACT)-based group therapy compared to individual ACT-therapy for adult cancer patients suffering from psychological distress. Participants will be recruited from referrals to the Cancer Rehabilitation Unit at Helsingborg Hospital, Sweden. A total number of 12-20 participants will be assigned to either the experimental group, receiving ACT group therapy, or the Active Control group, receiving individual ACT therapy. Both therapy interventions aim at increasing psychological flexibility. Sociodemographic as well as Medical information regarding their somatic disease will be collected at baseline assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Able to speak and understand the Swedish language
* Cancer patients at hospitals in Skånevård Sund (geographical area)
* Experience of psychological distress related to cancer diagnosis or cancer treatment
* Stable and planned cancer treatment or no ongoing treatment

Exclusion Criteria:

* Severe cognitive problems
* Severe psychiatric disorder
* Ongoing substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Swedish Acceptance and Action Questionnaire (SAAQ) | Baseline and end of treatment (baseline+3-16 weeks)
  Measures self-reported psychological flexibility on a 7-point likert scale. The questionnaire includes a total of 6 items. Each item is scored 1-7 (1=never true, 7=always true), yielding a total between 7 and 42 where a higher number indicates lower psychological flexibility.

SECONDARY OUTCOMES:
Change in Swedish Acceptance and Action Questionnaire (SAAQ) | Baseline and follow up (6 weeks after end of treatment)
  Measures self-reported psychological flexibility on a 7-point likert scale. The questionnaire includes a total of 6 items. Each item is scored 1-7 (1=never true, 7=always true), yielding a total between 7 and 42 where a higher number indicates lower psychological flexibility.
Change in Swedish Acceptance and Action Questionnaire (SAAQ) | End of treatment (baseline + 3-16 weeks) and follow up (6 weeks after end of treatment)
  Measures self-reported psychological flexibility on a 7-point likert scale. The questionnaire includes a total of 6 items. Each item is scored 1-7 (1=never true, 7=always true), yielding a total between 7 and 42 where a higher number indicates lower psychological flexibility.
Change in Generalized Anxiety Disorder 7 (GAD-7) | Baseline and end of treatment (baseline+3-16 weeks)
  Measures self-reported severity and frequency of symptoms of generalized anxiety disorder over the last 2 weeks on a 4-point likert scale. The questionnaire includes a total of 7 items. Each item is scored from 0-3 (0=never, 3=daily), yielding a total between 0 and 21 where a higher number indicates a higher severity of the patient's anxiety.
Change in Generalized Anxiety Disorder 7 (GAD-7) | Baseline and follow up (6 weeks after end of treatment)
  Measures self-reported severity and frequency of symptoms of generalized anxiety disorder over the last 2 weeks on a 4-point likert scale. The questionnaire includes a total of 7 items. Each item is scored from 0-3 (0=never, 3=daily), yielding a total between 0 and 21 where a higher number indicates a higher severity of the patient's anxiety.
Change in Generalized Anxiety Disorder 7 (GAD-7) | End of treatment (baseline+3-16 weeks) and follow up (6 weeks after end of treatment)
  Measures self-reported severity and frequency of symptoms of generalized anxiety disorder over the last 2 weeks on a 4-point likert scale. The questionnaire includes a total of 7 items. Each item is scored from 0-3 (0=never, 3=daily), yielding a total between 0 and 21 where a higher number indicates a higher severity of the patient's anxiety.
Change in Patient Health Questionnaire 9 (PHQ-9) | End of treatment (baseline+3-16 weeks) and follow-up (6 weeks after end of treatment)
  Measures self-reported presence and severity of symptoms of depression over the last 2 weeks on a 4-point likert scale. The questionnaire includes a total of 9 items. Each item is scored from 0-3 (0=not at all, 3=nearly every day), yielding a total between 0 and 27 where a higher number indicates more severe symptoms of depression.
Change in Patient Health Questionnaire 9 (PHQ-9) | Baseline and follow-up (6 weeks after end of treatment)
  Measures self-reported presence and severity of symptoms of depression over the last 2 weeks on a 4-point likert scale. The questionnaire includes a total of 9 items. Each item is scored from 0-3 (0=not at all, 3=nearly every day), yielding a total between 0 and 27 where a higher number indicates more severe symptoms of depression.
Change in Patient Health Questionnaire 9 (PHQ-9) | Baseline and end of treatment (baseline + 3-16 weeks)
  Measures self-reported presence and severity of symptoms of depression over the last 2 weeks on a 4-point likert scale. The questionnaire includes a total of 9 items. Each item is scored from 0-3 (0=not at all, 3=nearly every day), yielding a total between 0 and 27 where a higher number indicates more severe symptoms of depression.
Change in RAND 36-item Health Survey (RAND-36) | Baseline and end of treatment (baseline + 3-16 weeks)
  Measures self-reported health related quality of life. The questionnaire includes a total of 35 items within 8 subscales (physical function, physical role-function, emotional role-function, social function, psychological well-bering, vitality, pain and general health). For each scale, using the standardised score calculation, a scale score is given between 0 and 100, where 0 is worse and 100 is best.
Change in RAND 36-item Health Survey (RAND-36) | Baseline and follow up (6 weeks after end of treatment)
  Measures self-reported health related quality of life. The questionnaire includes a total of 35 items within 8 subscales (physical function, physical role-function, emotional role-function, social function, psychological well-bering, vitality, pain and general health). For each scale, using the standardised score calculation, a scale score is given between 0 and 100, where 0 is worse and 100 is best.
Change in RAND 36-item Health Survey (RAND-36) | End of treatment (baseline+3-16 weeks) and follow-up (6 weeks after end of treatment)
  Measures self-reported health related quality of life. The questionnaire includes a total of 35 items within 8 subscales (physical function, physical role-function, emotional role-function, social function, psychological well-bering, vitality, pain and general health). For each scale, using the standardised score calculation, a scale score is given between 0 and 100, where 0 is worse and 100 is best.

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Nystrom, PhD, Principal Investigator — Region Skane
Locations (1):
- Cancerrehabiliteringsmottagningen Helsingborg, Helsingborg, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No